

Research Evaluating Sports ConcUssion Events -

Rapid Assessment of Concussion and Evidence for Return

Informed Consent document dates: CArBON and CARS (28th August 2018)

IRAS ID: 231314





## Consent form

**Title of Project:** Competitor Assessment at Baseline; Ocular and Neuroscientific (CArBON)

Name of study team member present:

| The study team consists of individuals associated with the RESCUE-RACER programme working a | at |
|---|---|
| Cambridge University Hospitals Trust and/or the University of Cambridge. | Ple |

ease initial box 1. I confirm that I have read the information sheet dated ...... (version......) for the **CArBON** study. I have had the opportunity to consider the information, ask questions and have had these answered to my satisfaction. 2. I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. 3. I understand that the information collected about me will be used to support other research in the future and may be shared anonymously with other researchers in the UK and abroad. 4. I understand that anonymised study results will likely be presented to the scientific community (including publication and presentation). Please answer YES/NO 5. I understand that relevant sections of my motorsport records may be looked at by members of the study team (including medical notes, previous concussion assessments and accident data). I give permission for these individuals to access my records.

6. I understand that relevant sections of my medical notes may be looked at by members of study team, or from regulatory authorities where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records, including contact with my GP.

IRAS ID: 231314





| | | | Please answer<br>YES/NO |
|---|---|---|---|
| 7. I agree that <u>anonymised</u> future ethically approved | | during the <b>CArBON</b> study may be use | Please initial box |
| 8. I agree to take part in the <b>CArBON</b> study. | | | |
| 9. I agree not to participate | in any driving activity unt | il 1 hour after OVRT testing. | |
| Name of Participant (please print) | Signature | <br>Date | |
| If participant is aged less than | 18 years <u>;</u> | | |
| Name of Parent/Guardian (please print) | Signature | Date | |
| Name of Study team member (please print) | Signature | <br>Date | |

Two copies are required: research file, participant





## Consent form

**Title of Project:** Concussion Assessment and Return to motorSport (CARS)

| Name of study team member present: | |
|---|---|
| The study team consists of individuals associated with the <b>RESCUE-RACER</b> programme working at Cambridge University Hospitals Trust and/or the University of Cambridge. Ple | ase initial<br>box |
| 10. I confirm that I have read the information sheet dated (version) for the <b>CARS</b> study. I have had the opportunity to consider the information, ask questions and have had these answered to my satisfaction. | |
| 11. I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | |
| 12. I understand that the information collected about me will be used to support other research in the future and may be shared anonymously with other researchers in the UK and abroad. | |
| 13. I understand that anonymised study results will likely be presented to the scientific community (including publication and presentation). | |
| | se answer<br>/ES/NO |
| 14. I understand that relevant sections of my motorsport records may be looked at by members of<br>the study team (including medical notes, previous concussion assessments and accident data). I give permission for these individuals to access my records. | |
| 15. I understand that relevant sections of my medical notes may be looked at by members of study team, or from regulatory authorities where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records, including contact with my GP. | |

IRAS ID: 231314





Please answer

| | | | YES/NO |
|---|---|---|---|
| 16. I agree that <u>anonymised</u> dar<br>future ethically approved stu | | ring the CARS study may be used for | Please initial |
| 17. I agree to take part in the C | ARS study. | | box |
| 18. I agree not to participate in | any driving activity until 1 | hour after OVRT testing. | |
| | | | - |
| Name of Participant<br>(please print) | Signature | Date | |
| f participant is aged less than 18 | 3 years; | | |
| | | | - |
| Name of Parent/Guardian<br>(please print) | Signature | Date | |
| Name of Study team member (please print) | Signature | <br>Date | - |
| Two copies are required: researd | ch file, participant | | |